CLINICAL TRIAL: NCT00007839
Title: Phase I/II Study to Assess the Safety and Efficacy of Low Doses of Beta LT in Patients With B-Cell Lymphoma
Brief Title: Beta Alethine in Treating Patients With Low-Grade Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LifeTime Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068279; LIFETIME-LTP-99-02; LIFETIME-IRB-0300202; NCI-V00-1628
Record Dates: First submitted 2001-01-06; First posted 2003-10-08 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2010-04

CONDITIONS: Lymphoma
Keywords: stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — alethine

INTERVENTIONS:
Drug: beta alethine

SUMMARY:
RATIONALE: Biological therapies such as beta alethine use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I/II trial to study the effectiveness of beta alethine in treating patients who have low-grade lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor effects of low-dose beta-alethine in patients with low grade B-cell lymphoma.
* Assess the effects of this regimen on delayed-type hypersensitivity in these patients.
* Assess the safety of this regimen in this patient population.

OUTLINE: This is an multicenter study.

Patients receive low-dose beta-alethine subcutaneously once every 2 weeks for a total of 6 doses in the absence of unacceptable toxicity. Patients with no evidence of tumor progression may receive additional courses of therapy.

Patients are followed for 2 weeks from the last dose or for a minimum of 30 days if they withdraw due to an adverse event.

PROJECTED ACCRUAL: Approximately 13-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low grade B-cell lymphoma

  * Measurable residual disease after maximal response to prior chemotherapy OR
  * Indolent disease not yet requiring therapy
* No congenital immunodeficiency associated lymphoma
* No primary lymphoma of the brain
* No active brain involvement or leptomeningeal disease NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* At least 4 months

Hematopoietic:

* Neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT/SGPT no greater than 2.5 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 2.0 mg/dL
* Calculated creatinine clearance at least 60 mL/min

Cardiovascular:

* No uncontrolled angina, heart failure, or arrhythmia
* No acute changes on EKG

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No AIDS
* Adequate nutritional status (total protein at least 60.0 g/L)
* No active bacterial infections (e.g., abscess or with fistula)
* No nonmalignant disease that would preclude study
* No history of alcoholism, drug addiction, or psychotic disorders that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior bone marrow transplantation allowed
* At least 4 weeks since prior immunotherapy or cytokines

Chemotherapy:

* See Disease Characteristics
* Prior intensive chemotherapy with stem cell support allowed
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or high dose carboplatin)

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy to more than 25% of bone marrow

Surgery:

* Recovered from prior surgery
* No prior solid organ transplantation

Other:

* No concurrent antiinflammatory agents including aspirin, or over the counter or prescription nonsteroidal antiinflammatory drugs
* No concurrent immunosuppressive agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Suzin Mayerson, PhD, Study Chair — LifeTime Pharmaceuticals
Locations (1):
- Victory Over Cancer, Rockville, Maryland, United States